CLINICAL TRIAL: NCT00005931
Title: A Multicenter, Open-Label, Phase II Study of SU5416 in Patients With Therapy-Refractory Cutaneous AIDS-Related Kaposi's Sarcoma
Brief Title: SU5416 in Patients With AIDS-Related Kaposi's Sarcoma Who Have Not Responded to Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SUGEN (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 310B; SU5416.027
Record Dates: First submitted 2000-06-30; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2000-12

CONDITIONS: Sarcoma, Kaposi; HIV Infections
Keywords: Skin Neoplasms; Sarcoma, Kaposi; Acquired Immunodeficiency Syndrome; Antineoplastic Agents; Enzyme Inhibitors; SU 5416; Protein-Tyrosine Kinase
MeSH Terms: conditions — Sarcoma, Kaposi; HIV Infections; Skin Neoplasms; Acquired Immunodeficiency Syndrome | interventions — Semaxinib

INTERVENTIONS:
Drug: SU5416

SUMMARY:
The purpose of this study is to test the effectiveness of SU5416 in patients with AIDS-related Kaposi's sarcoma (KS).

DETAILED DESCRIPTION:
Patients are given SU5416 via twice-weekly intravenous infusions in 4-week treatment cycles. Any patient who has not experienced unacceptable toxicity and who is deemed to be responding to the study drug (no evidence of disease progression) is permitted to continue receiving SU5416 in 4-week treatment cycles (up to a maximum of 1 year of therapy) until that patient experiences either unacceptable toxicity or tumor progression, as defined in the protocol.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are at least 18 years old.
* Have KS.
* Have taken paclitaxel, DaunoXome, or Doxil for KS and they have either not gotten better or could not tolerate treatment therapy.
* Have 1 of the following symptoms for KS: 5 lesions (sores), generalized KS-related edema (swelling) without sores, or KS-related edema of the arms and legs.
* Agree to use an effective method of birth control during the study.

Exclusion Criteria

Patients will not be eligible for this study if they:

* Are pregnant or breast-feeding.
* Are allergic to Cremophor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30

CONTACTS AND LOCATIONS:
Locations (1):
- Alison L. Hannah, South San Francisco, California, United States